CLINICAL TRIAL: NCT02624596
Title: NMDAR Modulation As a Therapeutic Target and Probe of Neural Dysfunction in OCD
Brief Title: Understanding How Ketamine Brings About Rapid Improvement in OCD
Acronym: MKET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 34622
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): OCD patients in this arm will receive 0.5mg/kg of ketamine - one single infusion
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): OCD patients in this arm will receive 0.045mg/kg of midazolam - one single infusion
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — OCD patients in this arm will receive 0.5mg/kg of ketamine - one single infusion
  Other Names: Ketamine Hydrochloride
  Arms: Ketamine
Drug: Midazolam — OCD patients in this arm will receive 0.045mg/kg of midazolam - one single infusion
  Other Names: Midazolam Hydrochloride
  Arms: Midazolam

SUMMARY:
The purpose of this study is to understand how ketamine brings about rapid improvement in Obsessive-Compulsive Disorder (OCD) symptoms.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a chronic and disabling disorder that costs the economy over $2 billion annually and represents a significant public health problem. This study aims to build on our discovery that a potent NMDA receptor antagonist, ketamine, has rapid (in hours) and robust therapeutic effects in OCD. The proposed projects test the acute mechanism of action of ketamine at the level of molecules, circuits, and network synchrony to determine how NMDA receptor antagonism modifies the underlying pathology of OCD to relieve repetitive thoughts and behaviors.

ELIGIBILITY:
Inclusion Criteria for participants with OCD:

* age 18-65
* Primary diagnosis of OCD
* Sufficient severity of OCD symptoms
* ability to tolerate a treatment-free period
* capacity to provide informed consent

Inclusion criteria for healthy controls:

* ages 18-65
* capacity to provide informed consent

Exclusion criteria for participants with OCD:

* Psychiatric or medical conditions that make participation unsafe
* pregnant or nursing females
* concurrent use of any medications that might increase the risk of participation (e.g. drug interactions)
* presence of metallic device or dental braces

Exclusion criteria for healthy controls:

* any current or lifetime psychiatric diagnosis
* pregnant or nursing females
* major medical or neurological problem
* presence of metallic device or dental braces

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
improvement in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Up to 6 months
  Improvement in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.

SECONDARY OUTCOMES:
Regional gamma-aminobutyric acid, glutamate/glutamine levels derived from 3T Magnetic Resonance Spectroscopy | up to 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Bandeira ID, Lins-Silva DH, Cavenaghi VB, Dorea-Bandeira I, Faria-Guimaraes D, Barouh JL, Jesus-Nunes AP, Beanes G, Souza LS, Leal GC, Sanacora G, Miguel EC, Sampaio AS, Quarantini LC. Ketamine in the Treatment of Obsessive-Compulsive Disorder: A Systematic Review. Harv Rev Psychiatry. 2022 Mar-Apr 01;30(2):135-145. doi: 10.1097/HRP.0000000000000330. PMID 35267254
- See also: Stanford Medicine Faculty Page — https://med.stanford.edu/profiles/carolyn-rodriguez?tab=bio
- See also: Rodriguez Lab Website — https://med.stanford.edu/rodriguezlab/research.html